CLINICAL TRIAL: NCT06118255
Title: Open-Label, Single-Arm, Phase 3 Study to Evaluate Safety, Tolerability, and Pharmacokinetics of Fenfluramine (Hydrochloride) in Infants 1 Year to Less Than 2 Years of Age With Dravet Syndrome
Brief Title: A Study to Evaluate Safety, Tolerability, and Pharmacokinetics of Fenfluramine (Hydrochloride) in Infants 1 Year to Less Than 2 Years of Age With Dravet Syndrome
Acronym: ORCHID
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: UCB BIOSCIENCES, Inc. (Industry)
Responsible Party: Sponsor
Organization: UCB Pharma (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EP0213; 2022-502359-75 (Registry Identifier: EU Clinical Trials); U1111-1289-2867 (Other: World Health Organization (WHO))
Record Dates: First submitted 2023-10-23; First posted 2023-11-07 (Actual); Last update posted 2025-12-17 (Actual); Status verified 2025-12

CONDITIONS: Dravet Syndrome
Keywords: Dravet syndrome; pediatrics; Fintepla; fenfluramine
MeSH Terms: conditions — Epilepsies, Myoclonic | interventions — Fenfluramine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Fenfluramine Open-label (Experimental): All study participants will initiate fenfluramine hydrochloride (HCl) treatment at 0.2 mg/kg/day in the Dose-Finding Period and may be up-titrated to a maximum of 0.8 mg/kg/day based on the Investigators discretion. The dose of fenfluramine HCl can be flexibly titrated during the Maintenance Period. Study participants, who discontinue early will participate in the Taper Period. All participants will complete an End of Treatment (EOT) Visit.
  Interventions: Drug: fenfluramine

INTERVENTIONS:
Drug: fenfluramine — The study drug, fenfluramine HCl, is an oral solution to be administered in equal doses twice daily (BID). It will be based on the current dose and participant's weight (kg).
  Other Names: Fintepla

SUMMARY:
The primary purpose of this study is evaluate the safety and tolerability of fenfluramine hydrochloride (HCl) 0.2 to 0.8 mg/kg/day in infants 1 year to less than 2 years of age with Dravet syndrome.

ELIGIBILITY:
Inclusion Criteria:

* Participant is ≥1 to <2 years of age as of the day of the first administration of study drug
* Participant has a documented diagnosis or likely diagnosis of Dravet syndrome according to the International League Against Epilepsy (ILAE) criteria and as agreed by the Epilepsy Study Consortium (ESC)
* Participant must be currently receiving ≥1 concomitant anti seizure medication (ASM) at a stable dose for ≥4 weeks prior to the Screening Visit and is expected to remain stable throughout the study. Rescue medications for seizures are not counted towards the total number of ASMs
* Participant must have drug resistant epilepsy as defined as a history of failure of adequate trials of 2 tolerated, appropriately chosen and used antiepileptic drug schedules (whether as monotherapies or in combination) to achieve sustained seizure freedom
* Participants must have ≥1 countable motor seizures (CMS) during the Baseline Period. The CMS include distinct seizures of generalized tonic-clonic, bilateral clonic, focal motor, bilateral tonic, atonic (drop), bilateral tonic/atonic, or focal to bilateral tonic-clonic type. If the participant fails to have ≥1 qualifying seizures in 28 days, the Baseline Period may be extended by an additional 14 days with Sponsor approval. Participants with an extended Baseline Period must still have ≥1 CMS in the 28 days immediately prior to the day of the first administration of study drug
* Body weight is ≥8 kg
* Males and females

Exclusion Criteria:

* Participant has a known hypersensitivity to fenfluramine hydrochloride (HCl) or any of the excipients in the study drug
* Participant has an exclusionary cardiovascular or cardiopulmonary abnormality based on echocardiogram (ECHO), electrocardiogram (ECG), or physical examination and is not approved for entry by the central cardiac reader
* Participant has a diagnosis of pulmonary arterial hypertension
* Participant has a clinically significant medical condition, including chronic obstructive pulmonary disease, interstitial lung disease, or portal hypertension, or has had clinically relevant symptoms or a clinically significant illness currently or in the 4 weeks prior to the Screening Visit, other than epilepsy, that in the opinion of the Investigator would negatively impact study participation, collection of study data, or pose a risk to the participant
* Participant has current or past history of cardiovascular or cerebrovascular disease, such as cardiac valvulopathy, myocardial infarction or stroke, severe ventricular arrhythmias, or clinically significant structural cardiac abnormality, including but not limited to mitral valve prolapse, atrial or ventricular septal defects, patent ductus arteriosus, and patent foramen ovale with reversal of shunt. (Note: Patent foramen ovale or a bicuspid aortic valve are not considered exclusionary.)
* Participant has a current or past history of glaucoma
* Participant has moderate to severe hepatic impairment, assessed based on the Child-Pugh classification system
* Participant has moderate to severe renal impairment (estimated glomerular filtration rate <50 mL/min/1.73 m^2 calculated with the updated Bedside Schwartz equation for children
* QT interval corrected (QTc) >450 msec
* Participant is taking >4 concomitant ASMs
* Participant is receiving concomitant treatment with cannabidiol other than Epidiolex/Epidyolex or is being actively treated with tetrahydrocannabinol (THC) or any marijuana product for any condition
* Participant is receiving concomitant therapy with any of the following: centrally-acting anorectic agents; monoamine-oxidase inhibitors; any centrally-acting compound with clinically appreciable amount of serotonin agonist or antagonist properties, including serotonin reuptake inhibition; other centrally-acting noradrenergic agonists, including atomoxetine; or cyproheptadine. Disallowed medications are subject to washout of ≥5 half-lives before the first day of study drug administration
* Participant is currently receiving another investigational product(s) or has received another investigational product within 30 days or within <5 times the half-life of that investigational product, whichever is longer, prior to the Screening Visit
* Participant has previously been treated with Fintepla (fenfluramine HCl) prior to the Screening Visit

Ages: 1 Year to 23 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 25 (Actual)
Dates: Start 2024-05-21 (Actual); Primary Completion 2026-09-03 (Estimated); Study Completion 2026-11-20 (Estimated)

PRIMARY OUTCOMES:
Change from Baseline in QT interval corrected by Fridericia (QTcF) at Visit 13 (End of Treatment/Early Termination (EOT/ET)) | Week 52 (Visit 13; EOT/ET), compared to Baseline
  QTcF is the QT interval corrected for heart rate according to Fridericia's formula. Higher values correspond to prolongation of QT interval.
Occurrence of a treatment-emergent (ie, post-Baseline through Visit 13 [EOT/ET]) result which meets the FDA case definition of drug associated valvulopathy | From post-Baseline (Day 1) through Visit 13 (EOT/ET) (up to 52 weeks)
  Drug associated valvulopathy refers to aortic regurgitation with severity mild or greater and/or mitral regurgitation with severity moderate or greater.
Occurrence of treatment-emergent (ie, post-Baseline through Visit 13 [EOT/ET]) clinically confirmed valvular heart disease (VHD) | From post-Baseline (Day 1) through Visit 13 (EOT/ET) (up to 52 weeks)
  Clinically confirmed VHD is an aortic regurgitation with mild or greater severity and/or a mitral regurgitation with moderate or greater severity.
Change from Baseline in body weight (Z-score) at each visit | Week 1 (Visit 3), Week 4 (Visit 5), Week 8 (Visit 7), Week 12 (Visit 8), Week 16 (Visit 9), Week 20 (Visit 10), Week 26 (Visit 11), Week 39 (Visit 12), Week 52 (Visit 13), Postdose Safety Follow-Up (Visit 14), compared to Baseline
  Body weight (Z-score) refers to the number of standard deviations a participant's body weight lies from the mean, when compared to others of similar gender and age.
Change from Baseline in recumbent length (Z-score) at each visit | Week 1 (Visit 3), Week 4 (Visit 5), Week 8 (Visit 7), Week 12 (Visit 8), Week 16 (Visit 9), Week 20 (Visit 10), Week 26 (Visit 11), Week 39 (Visit 12), Week 52 (Visit 13), Postdose Safety Follow-Up (Visit 14), compared to Baseline
  Recumbent length (Z-score) refers to the number of standard deviations a participant's body weight lies from the mean, when compared to others of similar gender and age.
Occurrence of a clinically significant abnormality on the neurological examination at each visit | Week 1 (Visit 3), Week 4 (Visit 5), Week 8 (Visit 7), Week 12 (Visit 8), Week 16 (Visit 9), Week 20 (Visit 10), Week 26 (Visit 11), Week 39 (Visit 12), Week 52 (Visit 13), Postdose Safety Follow-Up (Visit 14), compared to Baseline
  A complete neurological examination will be conducted by the investigator for each participant covering cranial nerves, muscle strength and tone, reflexes, coordination, sensory function, and gait.

SECONDARY OUTCOMES:
Percentage change from the Baseline Period (ie, Baseline) in monthly (28 days) countable motor seizure frequency (CMSF), during Weeks 9 through 20 | During Weeks 9 to 20, compared to Baseline
  The percentage change from the Baseline Period (Baseline) in "monthly (28 days) countable motor seizure frequency," or CMSF, during Weeks 9 through 20
Percentage change from Baseline in CMSF during Weeks 1 through 20 | During Weeks 1 to 20, compared to Baseline
  The percentage change from the Baseline Period (Baseline) in "monthly (28 days) countable motor seizure frequency," or CMSF, during Weeks 1 through 20
Percentage change from Baseline in CMSF during the Treatment Period (Week 1 through the EOT/ET Visit) | During the Treatment Period (Week 1 through EOT/ET) (up to 52 weeks), compared to Baseline
  The percentage change from the Baseline Period (Baseline) in "monthly (28 days) countable motor seizure frequency," or CMSF, during the Treatment Period (Week 1 through the EOT/ET Visit; up to 52 weeks)
Achievement of a Clinical Global Impression - Improvement (CGI-I) rating of "much improved" or "very much improved" as assessed by the Principal Investigator at Week 20 | At Week 20
  The CGI-I rating scale permits a global evaluation of the participant's improvement over time by the investigator on a 7-point scale.
Achievement of a CGI-I rating of "much improved" or "very much improved" as assessed by the parent/caregiver at Week 20 | At Week 20
  The CGI-I rating scale permits a global evaluation of the participant's improvement over time by the parent/caregiver on a 7-point scale.
Steady-state maximum plasma concentration (Cmax) of fenfluramine and norfenfluramine at Week 12 | At Week 12
  Mean peak (maximum) plasma concentration of fenfluramine and norfenfluramine will be reported at Study Week 12 when participants are in the Maintenance Period.
Steady-state minimum plasma concentration (Cmin) of fenfluramine and norfenfluramine at Week 12 | At Week 12
  Mean minimum plasma concentration of fenfluramine and norfenfluramine will be reported at Study Week 12 when participants are in the Maintenance Period.
Area under the plasma concentration time curve from time zero to 24 hours (AUC0 24) for steady-state fenfluramine and norfenfluramine at Week 12 | At Week 12
  Mean AUC0-24 values of fenfluramine and norfenfluramine will be reported at Study Week 12 when participants are in the Maintenance Period.

CONTACTS AND LOCATIONS:
Overall Officials: UCB Cares, Study Director — 001 844 599 2273
Locations (12):
- United States (3):
  - Ep0213 105, Memphis, Tennessee
  - Ep0213 107, Dallas, Texas
  - Ep0213 103, Seattle, Washington
- Belgium (2):
  - Ep0213 502, Brussels
  - Ep0213 501, Edegem
- Ep0213 303, Bielefeld, Germany
- Italy (4):
  - Ep0213 202, Florence
  - Ep0213 203, Genova
  - Ep0213 201, Roma
  - Ep0213 204, Roma
- United Kingdom (2):
  - Ep0213 403, Glasgow
  - Ep0213 401, London

IPD SHARING:
Plan to Share IPD: Yes
Data from this study may be requested by qualified researchers six months after product approval in the US and/or Europe, or global development is discontinued, and 18 months after trial completion. Investigators may request access to anonymized IPD and redacted study documents which may include: raw datasets, analysis-ready datasets, study protocol, blank case report form, annotated case report form, statistical analysis plan, dataset specifications, and clinical study report. Prior to use of the data, proposals need to be approved by an independent review panel at www.Vivli.org and a signed data sharing agreement will need to be executed. All documents are available in English only, for a pre-specified time, typically 12 months, on a password protected portal. This plan may change if a determination is made that the data cannot be adequately anonymized.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Data from this study may be requested by qualified researchers six months after product approval in the US and/or Europe or global development is discontinued, and 18 months after trial completion.
Access Criteria: Qualified researchers may request access to anonymized IPD and redacted study documents which may include: raw datasets, analysis-ready datasets, study protocol, blank case report form, annotated case report form, statistical analysis plan, dataset specifications, and clinical study report. Prior to use of the data, proposals need to be approved by an independent review panel at www.Vivli.org and a signed data sharing agreement will need to be executed. All documents are available in English only, for a pre-specified time, typically 12 months, on a password protected portal.
URL: https://vivli.org/